CLINICAL TRIAL: NCT02699801
Title: Dexmedetomidine Use in ICU Sedation and Postoperative Recovery in Elderly Patients and Post-cardiac Surgery
Acronym: DIRECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H15-02301
Record Dates: First submitted 2016-01-27; First posted 2016-03-04 (Estimated); Last update posted 2016-11-03 (Estimated); Status verified 2016-11

CONDITIONS: Delirium; Cognitive Decline; Post-operative Quality of Recovery
MeSH Terms: conditions — Delirium; Cognitive Dysfunction | interventions — Propofol; Dexmedetomidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Propofol (Active Comparator): Patients received propofol for post-operative sedation
  Interventions: Drug: propofol
- Dexmedetomidine (Active Comparator): Patients received dexmedetomidine for post-operative sedation
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: propofol — propofol for post-sternal closure sedation
  Arms: Propofol
Drug: Dexmedetomidine — dexmedetomidine for post-sternal closure sedation
  Arms: Dexmedetomidine

SUMMARY:
Increasing numbers of elderly patients are undergoing cardiac surgery. Elderly patients may have prolonged recovery following cardiac surgery when compared to other groups of patients, and are at higher risk of postoperative delirium, postoperative neurocognitive decline and reduced quality of life following hospital discharge.

The goals of sedation and analgesia for patients following cardiac surgery are multifold and include postoperative pain relief, the facilitation of ventilation, resolution of hypothermia and normalization of electrolyte balances. The choice of sedative agent however can impact postoperative outcomes. Dexmedetomidine has been associated with improved quality of recovery in patients undergoing major spine surgery and with a reduced incidence of delirium, both of which can impact a patient's quality of life following surgery. The investigators hypothesized that the use of dexmedetomidine as a sedative agent immediately following cardiac surgery in elderly patients would result in improved quality of recovery and a reduced incidence of delirium in the postoperative period, when compared to propofol. The investigators were also interested as to whether there was an associated improvement in neurocognitive outcomes in this population.

Questions:

* Does the use of dexmedetomidine as a sedative agent in ICU in elderly patients following cardiac surgery result in improved Quality of Recovery scores when compared with propofol?
* Does the use of dexmedetomidine as a sedative agent in ICU in elderly patients following CABG+/- AVR result in a reduced incidence of postoperative delirium as compared to propofol?
* Do these patients subsequently have a reduction in cognitive decline?

DETAILED DESCRIPTION:
Due to advances in surgical and anaesthetic techniques, increasing numbers of elderly patients are undergoing cardiac surgery. Elderly patients with multiple comorbidities undergoing cardiac surgery may have prolonged recovery following cardiac surgery when compared to other groups of patients, and are at higher risk of postoperative delirium, postoperative neurocognitive decline and reduced quality of life following hospital discharge.

Traditionally, outcomes following cardiac surgery were measured in terms of complication rates or mortality rates1. More recently however, quality of life (QoL) measures are increasingly being recognized as important outcome measurements following cardiac surgery2. Factors related to cardiac surgery and perioperative care which could potentially influence later QoL include quality of recovery following surgery, postoperative delirium, and postoperative neurocognitive decline.

Quality of recovery (QoR) is a newer concept, which aims to measure a patient's health status after surgery and anaesthesia. The use of dexmedetomidine during spinal surgery has been associated with improved quality of recovery in the early postoperative period3. There are suggestions that dexmedetomidine attenuates the increase in inflammatory mediators during a stress response4 which could have a role in the post-surgical stress response. There are no studies that have attempted to correlate dexmedetomidine use with quality of recovery following cardiac surgery.

The prevalence of delirium following cardiac surgery in patients over 60 years has been reported in the range 30-52% (5, 6). Delirium is a condition characterized by consciousness disturbances, concentration disorders, memory disturbances and hallucinations. There have been associations made between the choice of sedative and the prevalence of delirium in ICU patients. In a multicenter randomized trial predominantly involving medical patients in the ICU, those assigned to receive dexmedetomidine had a reduced risk of delirium and spent less time undergoing mechanical ventilation7. It is not known if the choice of sedation agent in this population impacts on the incidence of delirium following cardiac surgery. Delirium is associated with increased morbidity, prolonged hospital stay, increased mortality8

Cognitive decline refers to a condition in which intellectual abilities and memory seem impaired when the patient appears to have otherwise recovered from the surgery. It is a condition distinct from delirium or encephalopathy. Cognitive decline is common, and can be persist for months and years, following cardiac surgery. The reported incidence of cognitive decline after coronary artery bypass graft (CABG) has been reported as 53% at hospital discharge, 36% at 6 weeks and 42% at 5 years9. Elderly patient undergoing cardiac surgery are at increased risk for postoperative cognitive decline10. A strong relationship has been reported between cognitive decline and reduced quality of life following cardiac surgery11.

The goals of sedation and analgesia for patients following cardiac surgery are multifold and include postoperative pain relief, the facilitation of ventilation, resolution of hypothermia and normalization of electrolyte balances. The choice of sedative agent however can impact postoperative outcomes. Dexmedetomidine has been associated with improved quality of recovery in patients undergoing major spine surgery and with a reduced incidence of delirium, both of which can impact a patient's quality of life following surgery. We hypothesized that the use of dexmedetomidine as a sedative agent immediately following cardiac surgery in elderly patients would result in improved quality of recovery and a reduced incidence of delirium in the postoperative period, when compared to propofol. We were also interested as to whether there was an associated improvement in neurocognitive outcomes in this population.

ELIGIBILITY:
Inclusion Criteria:

* adults over 75yrs undergoing on-pump CABG +/- AVR

Exclusion Criteria:

* Consent refusal
* Language barrier
* Allergy to study drugs
* Receiving other alpha 2 agonists
* Dementia [mild cognitive impairment can be included]

Ages: 75 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-10 (Estimated); Study Completion 2018-02 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery - 40 | Post Operative Day 3
  Questionnaire

SECONDARY OUTCOMES:
Minnesota Cognitive Acuity Screen | Post Operative Day 5 and 6 months post operatively
  Questionnaire
Quality of Life Score SF-36 | 6 months post operatively
  Questionnaire

OTHER OUTCOMES:
Other Secondary Outcomes - Number of Incidences of delirium | Up to 6 months post surgery date
  Number of Incidences of delirium
Other Secondary Outcomes - Number of delirious days | Up to 6 months post surgery date
  Number of delirious days
Other Secondary Outcomes - Time to extubation | Up to 6 months post surgery date
  Time to extubation
Other secondary outcomes - Time to being discharge-ready from ICU | Up to 6 months post surgery date
  Time to being discharge-ready from ICU
Other secondary outcome - Length of hospital stay | Up to 6 months post surgery date
  Length of hospital stay
other secondary outcomes - Hospital mortality rate | Up to 6 months post surgery date
  Hospital mortality rate
other secondary outcomes - Adverse events (hypotension, bradycardia, increased troponin, PONV) | Up to 6 months post surgery date
  Adverse events (hypotension, bradycardia, increased troponin, PONV)

CONTACTS AND LOCATIONS:
Overall Officials: Janette Brohan, Principal Investigator — UBC
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No